CLINICAL TRIAL: NCT00954928
Title: The Safety of Hand Surgery in the Anticoagulated Patient
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ryan Calfee, MD, Associate Professor of Orthopaedic Surgery, Washington University School of Medicine
Other Study IDs: 09-0567
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Hand Surgery
Keywords: hand; wrist; anticoagulation; surgery; patients on anticoagulant medication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anticoagulated patients: Those patients taking Coumadin, Plavix, Aspirin, Lovenox.
- Control patients: Those patients having hand or wrist surgery who do not take any anticoagulant medication.

SUMMARY:
If operating on the anticoagulated patient has been safe for one of the investigators' surgeons for the past 10 years then providing prospective data that substantiates this could prevent complications related to the discontinuation of anticoagulation for hand surgery patients in the future.

DETAILED DESCRIPTION:
All eligible patients will be offered study enrollment pre-operatively. Demographic data collected during clinical interaction that will be gathered for research purposes and will included patient height, weight, age, anticoagulant medication(s) used with dosage/duration of use, indication for anticoagulant medication, and current INR if on warfarin. Preoperative examination will include measures of 2 point discrimination in the digits, distance of the fingertips from the distal palmar crease upon flexion, and the patient-based outcome surveys that are to be collected after surgery (Quick DASH, SF-12, Visual Analog Scales pain/swelling). These patients will then undergo the appropriate surgical procedure without discontinuing their anticoagulant medication.

To ensure that patients are not being placed at increased risk, this study's protocol will not alter the surgical practices of the attending surgeons involved. Specifically, all surgeons perform their hand and wrist surgery under tourniquet control but differ in whether the tourniquet is deflated prior to wound closure. Each surgeon will be free to manage the tourniquet as they feel appropriate. The placement of would drains will remain at the discretion of the attending surgeon on a case-by-case basis.

Local anesthetics may be injected but none will be mixed with epinephrine.

Procedures: (if applicable) Obtaining pre-operative INR values when appropriate, and performing surgery while continuing anticoagulants is already standard care for one faculty member. All post-operative care except the completion of the Quick DASH and Short Form 12, and visual analog ratings is part of standard clinical care. Research questionnaires should take no more than 20 minutes to complete per visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Taking daily anti-coagulant medication
* Having hand or wrist surgery

Exclusion Criteria:

* Surgery proximal to wrist
* Pregnant females
* INR > 3.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years of age having hand surgery while on anti-coagulant medication. Control subjects undergoing hand and wrist surgery without anticoagulant medications will be enrolled if they are over 18 years of age and able to consent to research participation. Patients on Coumadin with INR values less than or equal to 3.5 will be eligible for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2009-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
postoperative hematoma | 2 week, 4 week

SECONDARY OUTCOMES:
2 point discrimination | 2 week, 4 week
patient rated pain | 2 week, 4 week
patient rated function | 2 week, 4 week
ecchymosis | 2week , 4 week
joint range of motion | 2 week, 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Calfee, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Lindsley RC. Perioperative management of systemic oral anticoagulants in patients having outpatient hand surgery. J Hand Surg Am. 2008 Sep;33(7):1205-7. doi: 10.1016/j.jhsa.2008.05.026. PMID 18762121